CLINICAL TRIAL: NCT06062277
Title: Colchicine in Circulating Inflammatory Markers After Stroke
Brief Title: COlchicine iN Circulating Inflammatory Markers After StrokE (CONCISE)
Acronym: CONCISE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College Dublin (Other)
Collaborators: Mater Misericordiae University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCRC/23/04
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Ischemic Stroke; Atherosclerosis
Keywords: hsCRP; ischaemic stroke; atherosclerosis
MeSH Terms: conditions — Ischemic Stroke; Atherosclerosis | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Before and after intervention paired cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm Study (Other): Paired cohort before and after study. Each participant will act as their own control.
  All participants will receive the intervention: study drug colchicine 0.5mg orally once daily for a treatment period of 30 days.
  Interventions: Drug: Colchicine 0.5 MG

INTERVENTIONS:
Drug: Colchicine 0.5 MG — one oral tablet daily for 30 days

SUMMARY:
The goal of this phase 2, before-and-after interventional study is to investigate the effect of colchicine treatment on serum biomarkers of inflammation in patients with a history of stroke and atherosclerosis.

Participants meeting inclusion criteria will have blood samples drawn at baseline, will be dispensed colchicine 0.5mg daily for a treatment period of 30 days and have blood samples drawn again at follow-up. All blood samples will be analysed for a panel of inflammatory blood markers and the change in blood inflammatory markers from baseline to end of treatment will be calculated.

DETAILED DESCRIPTION:
Patients with a history of stroke or TIA, atherosclerosis and hsCRP≥2mg/L at baseline will be eligible for inclusion. Participants ≥18 years and ≤90 years, with no race, ethnicity or sex exclusions will be recruited. The target sample size is 91 participants. The sample size was calculated based on a paired two-sided t-test, using a 33% effect size, setting alpha at 0.05 and power at 0.8, and allowing for up to 20% non-adherence with colchicine.

Participants will receive 30 days treatment with pleiotropic anti-inflammatory agent colchicine 0.5mg tablets orally once daily for 30 days. A panel of blood inflammatory markers will be drawn pre and post treatment. Outcomes will be the calculated change in blood inflammatory marker panel, including hsCRP and IL-6, comparing before treatment levels with after treatment levels. This is a before and after paired cohort study, each participant will act as their own control.

All participants will receive the intervention study medication, colchicine 0.5mg orally once daily. Medication adherence will be ascertained by pill count and tolerability assessed using the MAQ questionnaire. MAQ questionnaire is a 6 item questionnaire which will assess each participants perception of the convenience, taste, look and smell, effect, side-effects and overall acceptability of the study drug, colchicine, on a likert scale.

Baseline characteristics will be collected including participant demographics, past medical history, medication use, blood pressure, BMI. These assessments will be repeated at the follow-up visit. This information will be collected with participant consent via participant reported history, physical exam, office blood pressure and weight measurement, and with reference to medical notes.

ELIGIBILITY:
Inclusion Criteria:

1. Free of chronic kidney disease and eGFR>50ml/min on baseline blood tests
2. Serum hsCRP≥2mg/L measured during the screening phase or on routine bloods in the year prior to recruitment.
3. History of ischaemic stroke or TIA
4. presence of atheroma, including intracranial or extracranial atheroma causing ≥30% stenosis or occlusion ipsilateral to the infarct; any atheroma proximal to the infarct in patients with cryptogenic stroke or ESUS in whom an alternative mechanism is not felt to be more likely in the opinion of the physician; history of ischaemic heart disease, peripheral arterial disease or has undergone revascularisation procedures for either.

Exclusion Criteria:

1. Stroke or TIA likely caused by identified atrial fibrillation (permanent or paroxysmal)
2. Stroke or TIA caused by other identified cardiac source (intracardiac thrombus, endocarditis, metallic heart value, low ejection fraction <30%)
3. History of myalgia with raised CK on statin therapy
4. Blood dyscrasia (Hb <10g/dl; Plt <150x10^9/L; WCC <4x10^9/L) or other history of blood dyscrasia requiring follow-up with Haematology
5. Impaired hepatic function (transaminases >twice ULN)
6. Concurrent treatment with contra-indicated drugs: CYP3A4 inhibitors (e.g. clarithromycin, erythomycin, telithromycin, macrolides, ketoconazole, itraconazole, voriconazole, tolbutamide, ritonavir, atazanavir, indinavir, other HIV protease inhibitors, verapamil, diltiazem, quinidine, digoxin, disulfiram) or P-GP inhibitors (e.g. cyclosporine) at screening
7. Symptomatic peripheral neuropathy or progressive neuromuscular disease
8. Pre-existing inflammatory bowel disease, Crohn's disease, Ulcerative colitis or chronic diarrhoea
9. Pre-existing inflammatory condition, intercurrent infection or other indication for regular anti-inflammatory therapies, e.g. steroid, NSAIDs, immunosuppressants.
10. Requirement for colchicine therapy for acute gout or gout prevention or other rheumatological disorder.
11. Known sensitivity of allergy to colchicine.
12. Active malignancy or known Hepatitis B, C or HIV infection.
13. Dementia or cognitive impairment sufficient to impair independence in basic activities of daily living.
14. People of childbearing potential (Must be >24 months free of menstrual periods)
15. Patient concurrently enrolled in the CONVINCE trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in hsCRP level | 4 weeks
  Percentage change in hsCRP level

SECONDARY OUTCOMES:
Change in IL-6 level | 4 weeks
  Percentage change in IL-6 level
Change in TNF-alpha level | 4 weeks
  Percentage change in TNF-alpha level
Change in MCP-1 level | 4 weeks
  Percentage change in MCP-1 level

OTHER OUTCOMES:
Medication tolerability, adherence and acceptability | 4 weeks
  Assessed using MAQ questionnaire and pill count. The MAQ is a 6 item questionnaire which assesses the participants perception of convenience, taste, look and smell, effect, side effects, overall acceptability of the study drug on a likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Stroke Clinical Trials Network Ireland, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No